CLINICAL TRIAL: NCT01073553
Title: Prospective, Randomized, Open Label, Crossover Study to Compare the Bioavailability Between Optocef (Cephalexin 500 mg Capsules) From Bayer and Keflex (Cephalexin 250 mg Capsules) From Eli Lilly po in Healthy Subjects Using Equivalent Concentrations
Brief Title: Cross-over Study to Prove Bioequivalence Between Two Brands of Cefalexin Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Corporación Bonima S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14784
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Anti-Infective Agents
MeSH Terms: interventions — Cephalexin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Cephalexin capsules (Optocef, BAYO5448 )
- Arm 2 (Active Comparator)
  Interventions: Drug: Cephalexin capsules (Keflex)

INTERVENTIONS:
Drug: Cephalexin capsules (Optocef, BAYO5448 ) — Single dose of 500 mg (One 500 mg capsule)
  Arms: Arm 1
Drug: Cephalexin capsules (Keflex) — Single dose of 500 mg (Two 250 mg capsules)
  Arms: Arm 2

SUMMARY:
A single dose, two treatments (two cephalexin capsules brands), two sequences, cross-over design was used with a washout of 7 days between the two study periods. Treatment groups balanced with the same number of healthy volunteers who were randomly (in two strata: male and female) assigned to the study drug administration sequences.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers age between 18 and 55 years old with normal vital signs, electrocardiogram (ECG), blood chemistry, liver function profile and urinalysis

Exclusion Criteria:

* History of illnesses or any organic abnormalities that could affect the results of the study
* History of tobacco or alcohol abuse or regular use of recreational or therapeutic drugs
* Subjects that have taken any medication within 14 days or that are in an elimination period of less than 7 half-lives (whichever is longest) before study startup

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Least square estimator of average maximum plasmatic concentration (log transformed) | After two months
Least square estimator of area under the pharmacokinetic curve (log transformed) | After two months

SECONDARY OUTCOMES:
Time at which maximum concentration is reached | After two months
Area under the pharmacokinetic curve from time=0 to last blood sample | After two months
Clearance constant of plasmatic concentration of study drug | After two months
Half life of plasmatic concentration of study drug | After two months
Adverse events collection | Up to six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Morelia, Michoacán, Mexico